CLINICAL TRIAL: NCT04824976
Title: Effects of Blueberries on Symptoms and Underlying Mechanisms of Functional Gastrointestinal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brain-Gut Research Group (Other)
Collaborators: Aalborg University (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Clive H Wilder-Smith, MD, Dr, Brain-Gut Research Group
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-01
Record Dates: First submitted 2020-03-31; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Active Comparator): Freeze-dried pure blueberry powder
  Interventions: Dietary Supplement: Blueberry
- Placebo (Placebo Comparator): Maltodextrin powder.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry — freeze-dried Northern highbush blueberry powder twice daily 15g = 60kcal
  Arms: Blueberry
Dietary Supplement: Placebo — matched powder maltodextrin twice daily = 60kcal
  Arms: Placebo

SUMMARY:
There is extensive pre-clinical evidence for potential health effects of blueberries. These are related, but not exclusively due to their high polyphenol content. This translational, clinical, randomized, cross-over, double-blind, placebo-controlled study will investigate the effects of blueberries in freeze-dried powder form on gastrointestinal and extra-gastrointestinal symptoms and function, as well as specific potential underlying mechanisms, in patients with the overlapping functional gastrointestinal disorders, irritable bowel syndrome and functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Fifty-five successive male or female patients with Functional Gastrointestinal Disorders FGID) enrolled from our Gastroenterology Group Practice (GGP) in Bern, Switzerland, classified as having either Irritable Bowel Syndrome (IBS), Functional Dyspepsia (FD) or both according to Rome 4 criteria (Drossman et al 2016; Schmulson et al. 2017)
* Age between 18 and 50 years
* Body mass index 18.5-29.9 kg/m2
* European / Caucasian ethnicity
* Able to give informed consent in German as documented by signature

Exclusion Criteria:

* Evidence of clinically significant disease, as assessed by usual clinical practice (history, blood and stool tests, imaging and endoscopy, as clinically required) and by investigator.
* Colonoscopy, antibiotics or probiotics within 2 weeks before or during the study.
* Planned dietary modifications (including polyphenol-rich fruit or vegetable smoothies, drinks or diets) or initiation of new treatments during the study period, besides the study interventions.
* Inability or contraindications to undergo the investigated intervention
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) | before and after 6 weeks of each treatment arm
  Validated scale of GI symptoms

SECONDARY OUTCOMES:
Change in cognitive neurological function tests | before and after 6 weeks of each treatment arm
  Cambridge Cognition neurocognitive test battery (CANTAB)
Change in musculoskeletal symptoms | before and after 6 weeks of each treatment arm
  Validated Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) scores
Change in breath gas concentrations and symptoms scores during fructose breath testing | before and after 6 weeks of each treatment
  AUCs (areas under curve) of hydrogen, methane and symptom scores during fructose breath tests
Change in laboratory markers for advanced glycation end products, tight junction proteins | before and after 6 weeks of each treatment
  Validated biochemical markers of advanced glycation, tight junction protein quantification

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Group Practice / Brain-Gut Research Group, Bern, Switzerland